CLINICAL TRIAL: NCT01513473
Title: A 26-week, Multinational, Multi-centre, Open-Labelled, Randomised, Parallel, Efficacy and Safety Comparison of Insulin Degludec and Insulin Detemir in Children and Adolescents 1 to Less Than 18 Years With Type 1 Diabetes Mellitus on a Basal-bolus Regimen With Insulin Aspart as Bolus Insulin, Followed by a 26-week Extension Investigating Long Term Safety (BEGIN™: Young 1)
Brief Title: A Trial Investigating the Efficacy and Safety of Insulin Degludec in Children and Adolescents With Type 1 Diabetes Mellitus
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3561; 2011-003148-39 (EudraCT Number); P/44/2010 (Other: EMA (PDCO)); U1111-1122-4758 (Other: WHO)
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Degludec + Insulin Aspart (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- Insulin Detemir +Insulin Aspart (Experimental)
  Interventions: Drug: insulin detemir; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec — Injected subcutaneously (under the skin) once daily. Dose individually adjusted.
  Arms: Insulin Degludec + Insulin Aspart
Drug: insulin detemir — Injected subcutaneously (under the skin) once or twice daily. Dose individually adjusted.
  Arms: Insulin Detemir +Insulin Aspart
Drug: insulin aspart — Injected subcutaneously (under the skin) as mealtime bolus insulin. Dose individually adjusted.

SUMMARY:
This trial is conducted in Africa, Asia, Europe and the United States of America (USA).

The aim of this trial is to investigate the efficacy and safety of insulin degludec in children and adolescents with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, and child assent as age-appropriate, obtained before any trial-related activities (Trial-related activities are any procedure that would not have been performed during normal management of the subject). The parents or legal representative of the child must sign and date the Informed Consent Form according to local requirements. The child, if possible, parents or legal representative of the child must sign and date the Child Assent Form according to local requirements
* Male or female diagnosed with type 1 diabetes mellitus (T1DM) (based on clinical judgement and supported by laboratory analysis as per local guidelines)
* Ongoing daily treatment with insulin (any regimen) for at least 3 months prior to Visit 1 (screening). No OADs (oral anti-diabetic drugs) are allowed
* HbA1c (glycosylated haemoglobin) maximum 11%

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products
* Previous participation in this trial. Participation is defined as randomisation
* Girls who are pregnant, breastfeeding or intend to become pregnant
* Girls who have had menarche and are not using adequate contraceptive measures according to local requirements
* Known hypoglycaemic unawareness or recurrent severe hypoglycaemic events as judged by the Investigator (trial physician)
* More than 1 diabetic ketoacidosis requiring hospitalisation within the last 3 months prior to Visit 1
* Significant concomitant disease, except for conditions associated with type 1 diabetes mellitus, which in the Investigator's opinion could interfere with the trial
* The receipt of any investigational drug within 1 month prior to Visit 1

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2012-01-16 (Actual); Primary Completion 2013-07-30 (Actual); Study Completion 2013-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (75):
- United States (26):
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, New Haven, Connecticut
  - Novo Nordisk Investigational Site, Gainesville, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Maitland, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Akron, Ohio
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
- Bulgaria (2):
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Varna
- Finland (5):
  - Novo Nordisk Investigational Site, Espoo
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Mikkeli
  - Novo Nordisk Investigational Site, OYS
  - Novo Nordisk Investigational Site, Pori
- France (4):
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Rennes
  - Novo Nordisk Investigational Site, Toulouse
- Germany (4):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Münster
- Italy (3):
  - Novo Nordisk Investigational Site, Chieti
  - Novo Nordisk Investigational Site, Genova
  - Novo Nordisk Investigational Site, Roma
- Japan (14):
  - Novo Nordisk Investigational Site, Chuo-shi, Yamanashi
  - Novo Nordisk Investigational Site, Fukushima
  - Novo Nordisk Investigational Site, Iruma-gun, Saitama
  - Novo Nordisk Investigational Site, Kobe-shi, Hyogo
  - Novo Nordisk Investigational Site, Kochi-shi, Kochi
  - Novo Nordisk Investigational Site, Kumamoto-shi, Kumamoto
  - Novo Nordisk Investigational Site, Maebashi-shi, Gunma
  - Novo Nordisk Investigational Site, Musashino-shi, Tokyo
  - Novo Nordisk Investigational Site, Niigata-shi, Niigata
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Sendai-shi, Miyagi
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Toyonaka-city, Osaka
  - Novo Nordisk Investigational Site, Tsu-shi, Mie
- Netherlands (5):
  - Novo Nordisk Investigational Site, Almere Stad
  - Novo Nordisk Investigational Site, Amersfoort
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Nijmegen
  - Novo Nordisk Investigational Site, Rotterdam
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Russia (4):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
- South Africa (2):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Norwich
  - Novo Nordisk Investigational Site, Sheffield

REFERENCES:
- [Background] Thalange N, Deeb L, Klingensmith G, Franco DR, Bardtrum L, Tutkunkardas D, Danne T. The rate of hyperglycemia and ketosis with insulin degludec-based treatment compared with insulin detemir in pediatric patients with type 1 diabetes: An analysis of data from two randomized trials. Pediatr Diabetes. 2019 May;20(3):314-320. doi: 10.1111/pedi.12821. Epub 2019 Feb 10. PMID 30666772
- [Result] Thalange N, Deeb L, Iotova V, Kawamura T, Klingensmith G, Philotheou A, Silverstein J, Tumini S, Ocampo Francisco AM, Kinduryte O, Danne T. Insulin degludec in combination with bolus insulin aspart is safe and effective in children and adolescents with type 1 diabetes. Pediatr Diabetes. 2015 May;16(3):164-76. doi: 10.1111/pedi.12263. Epub 2015 Feb 12. PMID 25683037
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 72 sites in 12 countries as follows:
  Bulgaria (2), Finland (5), France (4), Germany (3), Italy (2), Japan (15), Netherlands (5), Republic of Macedonia (2), Russian Federation (6), South Africa (2), United Kingdom (4), United States (22)
Groups:
- IDeg + IAsp: Subjects from 1 to 18 years of age were randomised into treatment arms, IDeg OD as basal insulin and IAsp as mealtime bolus insulin for a period of 26 weeks followed by extension trial for a period of 26 weeks. IDeg was given once a day at approximately the same time of the day. Basal and bolus insulin titration was done according to the lowest pre-breakfast SMPG value measured on the three days prior to the visit/ phone contact for IDeg.
- IDet + IAsp: Subjects from 1 to 18 years of age were randomised into treatment arms, IDet OD as basal insulin and IAsp as mealtime bolus insulin for a period of 26 weeks followed by extension trial for a period of 26 weeks. IDet was given once a day at approximately the same time of the day. Basal and bolus insulin titration was done according to the lowest pre-breakfast SMPG value measured on the three days prior to the visit/ phone contact for IDet.
Period: Main Trial (26 Weeks)
Arm/Group | IDeg + IAsp | IDet + IAsp
Started | 174 | 176 (1 subject was randomised but withdrew before the drug exposure.)
Exposed | 174 | 175
Completed | 170 | 165
Not Completed | 4 | 11
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Unclassified | 0 | 2
Period: Extension Trial (26 Weeks)
Arm/Group | IDeg + IAsp | IDet + IAsp
Started | 152 (18 subjects did not consent to participate in the extension trial.) | 128 (37 subjects did not consent to participate in the extension trial.)
Completed | 151 | 122
Not Completed | 1 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis set (FAS) included all randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg + IAsp | IDet + IAsp | Total
Number analyzed (Participants) | 174 | 176 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 174 | 176 | 350
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 78 | 156
  Male | 96 | 98 | 194

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin) (%) at 26 Weeks (Analysed by Central Laboratory)
Description: Change from baseline in HbA1c (%) after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: Full Analysis Set (FAS) Included all randomised subjects. LOCF values are presented for this endpoint.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg + IAsp | IDet + IAsp
Number analyzed (Participants) | 174 | 176
percentage of glycosylated haemoglobin | -0.20 (0.95) | -0.31 (0.89)

2. Secondary Outcome: Change From Baseline in HbA1c (%) at 52 Weeks (Analysed by Central Laboratory)
Description: Change from baseline in HbA1c (%) after 52 weeks of treatments.
Time Frame: Week 0, week 52
Population: Full Analysis Set (FAS) Included all randomised subjects. LOCF values are presented for this endpoint.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg + IAsp | IDet + IAsp
Number analyzed (Participants) | 174 | 176
percentage of glycosylated haemoglobin | -0.27 (1.07) | -0.22 (1.03)

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FPG) at 26 Weeks (Analysed by Central Laboratory)
Description: Change from baseline in FPG after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: Full Analysis Set (FAS) Included all randomised subjects. LOCF values are presented for this endpoint. 338 subjects were considered, as 12 excluded from PP analysis set, 1 withdrawn, 11 subjects did not have a valid HbA1c measurements after 12 weeks. FPG samples were missing for 9 subjects.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg + IAsp | IDet + IAsp
Number analyzed (Participants) | 157 | 160
mmol/L | -0.67 (5.99) | 0.50 (8.37)

4. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FPG) at 52 Weeks (Analysed by Central Laboratory)
Description: Change from baseline in FPG after 52 weeks of treatment.
Time Frame: Week 0, week 52
Population: Full Analysis Set (FAS) Included all randomised subjects. LOCF values are presented for this endpoint. 338 subjects were considered, as 12 excluded from PP analysis set, 1 withdrawn, 11 subjects did not have a valid HbA1c measurements after 12 weeks.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg + IAsp | IDet + IAsp
Number analyzed (Participants) | 157 | 160
mmol/L | -1.29 (6.53) | 1.10 (8.24)

5. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: TEAE is defined as an event that has onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment.
Time Frame: After 26 weeks and 52 weeks of treatment
Population: Safety analysis set included all subjects receiving at least one dose of investigational product.
Measure: Number; unit: events
Arm/Group | IDeg + IAsp | IDet + IAsp
Number analyzed (Participants) | 174 | 175
events
  TEAEs -26 weeks | 810 | 761
  TEAEs -52 weeks | 1462 | 1266

6. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Number of hypoglycaemic episodes (severe episodes or episodes with plasma glucose (PG) below or equal to 3.9 mmol/L (70 mg/dL) with or without symptoms of hypoglycaemia) during the trial; nocturnal [11 p.m. - 7 a.m./23:00 - 07:00] and over the entire day (24 hours)
Time Frame: After 26 weeks and 52 weeks of treatment
Population: Safety analysis set included all subjects receiving at least one dose of investigational product.
Measure: Number; unit: episodes
Arm/Group | IDeg + IAsp | IDet + IAsp
Number analyzed (Participants) | 174 | 175
episodes
  26 weeks (entire day) | 11712 | 10991
  26 weeks (nocturnal) | 1261 | 1458
  52 weeks (entire day) | 21560 | 18373
  52 weeks (nocturnal) | 2336 | 2586

7. Secondary Outcome: Number of Self-measured Hyperglycaemia (Episodes of PG Above 11.1 mmol/L (200 mg/dL))
Description: Episodes of PG >11.1mmol/L (200mg/dL)
Time Frame: After 26 weeks and 52 weeks of treatment
Population: Safety analysis set included all subjects receiving at least one dose of investigational product.
Measure: Number; unit: episodes
Arm/Group | IDeg + IAsp | IDet + IAsp
Number analyzed (Participants) | 174 | 175
episodes
  26 weeks | 31264 | 31173
  52 weeks | 58679 | 52831

8. Secondary Outcome: Number of Episodes With Self Monitored Blood Ketones Above 1.5 mmol (Capillary Blood Ketone Measurement to be Performed if Self-measured Plasma Glucose (SMPG) Exceeds 14.0 mmol/l (250 mg/dL))
Description: Blood ketones > 1.5mmol/L (Capillary blood ketone measurement to be performed if SMPG exceeds 14.0mmol/L (250mg/dL) )after 26 and 52 weeks of treatment
Time Frame: After 26 weeks and 52 weeks of treatment
Population: Full Analysis Set (FAS) Included all randomised subjects
Measure: Number; unit: episodes
Arm/Group | IDeg + IAsp | IDet + IAsp
Number analyzed (Participants) | 174 | 175
episodes
  26 weeks | 44 | 86
  52 weeks | 109 | 161

9. Secondary Outcome: Steady-state Plasma Concentrations of Insulin Degludec and Insulin Detemir on Three Different Visits (Three Different Weeks) During the First 26 Weeks of Treatment
Description: Steady state plasma concentrations of insulin degludec and insulin detemir on three different visits (three different weeks) during the trial.
Time Frame: Between week 1 and week 26
Population: Full Analysis Set (FAS) Included all randomised subjects. 1 subject was excluded from the analysis in the IDet arm as he was withdrawn before exposure to trial drug.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | IDeg + IAsp | IDet + IAsp
Number analyzed (Participants) | 174 | 175
pmol/L
  week 2 | 4540.4 (3999.0) | 3972.2 (6721.8)
  week 12 | 4148.1 (3726.9) | 5430.1 (9067.7)
  week 26 | 4105.6 (3456.5) | 6377.0 (10930.6)

10. Secondary Outcome: Insulin Antibodies (Insulin Degludec Specific, Insulin Detemir Specific, Insulin Aspart Specific and Antibodies Cross-reacting to Human Insulin)
Description: Antibody measurements : the values presented are week 52 (LOCF). The measurement of insulin antibodies after 26 and 52 weeks of treatment was done to fulfil the requirement of monitoring the long term immunogenicity. The unit of measure is percentage bound/total (%B/T) for these antibodies. The Antibodies cross reacting to Human Insulin is abbreviated as X-reacting AB Hu Insulin below)
Time Frame: After 52 weeks of treatment
Population: Full Analysis Set (FAS) Included all randomised subjects. LOCF values are presented for this endpoint.
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | IDeg + IAsp | IDet + IAsp
Number analyzed (Participants) | 174 | 175
%B/T
  Insulin aspart specific antibodies | 1.1 (2.6) | 1.5 (2.3)
  Insulin Detemir specific antibodies | NA (NA) — The antibody analysis was for subjects taking insulin detemir only | 6.1 (6.5)
  Insulin Degludec specific antibodies | 0 (0.3) | NA (NA) — The antibody analysis was for subjects taking insulin degludec only
  X-reacting AB Hu Insulin | 17.2 (7.7) | 26.0 (19.3)

ADVERSE EVENTS:
Time Frame: Treatment emergent events (after first trial product administration and no later than 7 days after last trial product administration)
Description: Safety analysis set included all subjects receiving at least one dose of investigational product.
Arm/Group | IDeg + IAsp | IDet + IAsp
Serious Adverse Events (participants affected / at risk) | 18/174 | 16/175
Other Adverse Events (participants affected / at risk) | 146/174 | 143/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg + IAsp (N=174) | IDet + IAsp (N=175)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood ketone body increased (Investigations) | 1 (2) | 2 (4)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (7) | 2 (2)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 3 (4)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg + IAsp (N=174) | IDet + IAsp (N=175)
Ear pain (Ear and labyrinth disorders) | 10 (12) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 12 (16) | 8 (12)
Abdominal pain upper (Gastrointestinal disorders) | 28 (42) | 17 (30)
Diarrhoea (Gastrointestinal disorders) | 22 (26) | 17 (25)
Nausea (Gastrointestinal disorders) | 13 (18) | 9 (12)
Vomiting (Gastrointestinal disorders) | 26 (38) | 22 (35)
Pyrexia (General disorders) | 30 (59) | 28 (45)
Bronchitis (Infections and infestations) | 9 (10) | 8 (11)
Ear infection (Infections and infestations) | 9 (11) | 11 (11)
Gastroenteritis (Infections and infestations) | 15 (19) | 22 (25)
Gastroenteritis viral (Infections and infestations) | 10 (15) | 8 (13)
Influenza (Infections and infestations) | 16 (19) | 18 (21)
Nasopharyngitis (Infections and infestations) | 72 (177) | 67 (141)
Pharyngitis (Infections and infestations) | 6 (7) | 9 (13)
Rhinitis (Infections and infestations) | 12 (19) | 14 (23)
Sinusitis (Infections and infestations) | 9 (13) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 34 (56) | 24 (58)
Viral infection (Infections and infestations) | 6 (8) | 10 (18)
Blood ketone body increased (Investigations) | 31 (78) | 46 (131)
Hypoglycaemia (Metabolism and nutrition disorders) | 26 (62) | 17 (31)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (16) | 5 (5)
Headache (Nervous system disorders) | 46 (106) | 51 (121)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (52) | 28 (41)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 7 (13)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 29 (45) | 34 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of plans by any investigator to publish and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to Novo Nordisk before submission for comments. Comments will be given within four weeks from receipt of the planned communication.